CLINICAL TRIAL: NCT04201275
Title: A Single-center, Randomized, Double-blind, Parallel, Placebo-controlled, Multiple Consecutive Dose Study to Assess the Tolerability, Pharmacokinetics and Pharmacodynamics of HEC74647 in Subjects With Chronic Hepatitis C Virus Infection
Brief Title: The Tolerability, Pharmacokinetics and Pharmacodynamics Study of HEC74647 in HCV-infected Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sunshine Lake Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEC74647-P-02
Record Dates: First submitted 2019-12-13; First posted 2019-12-17 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort 1 (Experimental): up to HEC74647PA capsule 50 mg once daily for 3 days
  Interventions: Drug: HEC74647PA capsule
- Cohort 2 (Experimental): up to HEC74647PA capsule 100 mg once daily for 3 days
  Interventions: Drug: HEC74647PA capsule
- Cohort 3 (Experimental): up to HEC74647PA capsule 200 mg once daily for 3 days
  Interventions: Drug: HEC74647PA capsule
- Cohort 4 (Placebo Comparator): up to placebo once daily for 3 days
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HEC74647PA capsule — Capsule administered orally once daily
  Arms: Cohort 1; Cohort 2; Cohort 3
Drug: placebo — HEC74647PA capsule matching placebo administered orally once daily
  Arms: Cohort 4

SUMMARY:
The goal of this study is to assess the tolerability, pharmacokinetics and antiviral activity of HEC74647 in HCV treatment naïve subjects with genotypes 1-6.

DETAILED DESCRIPTION:
All subjects will be receive QD doses of HEC74647 or the matching placebo for 3 days to assess the the tolerability, pharmacokinetics and antiviral activity at specified time-points during the study.All subjects also will be monitored for up to 8 days post-dose to determine the persistence of viral mutations.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and sign the ICF voluntarily prior to initiate the study;
* Able to complete the study according to the protocol;
* Agree to use protocol defined precautions against pregnancy
* Body weight of male and female subject should be ≥50 kg and ≥45 kg respectively; Body Mass Index (BMI) is between 18 and 30 kg/m2, inclusive;
* HCV treatment-naïve adult subjects with GT1-6 HCV infection
* HCV RNA level ≥ 5 log10 IU/mL at screening
* FibroScan score within 6 months≤12.5 kPa or Liver biopsy results within 12 months proved Non-cirrhosis

Exclusion Criteria:

* Smokers, who smoke more than 5 cigarettes/day within 3 months before the study;
* Drink frequently, namely alcohol consumption are 14 units per week (1 unit = 285 mL of beer, or 25 mL of strong wine, or 100 mL of grape wine);
* Donated blood or massive blood loss within 3 months before screening (>450 mL）;
* Have any disease that increases the risk of bleeding, such as acute gastritis or stomach and duodenal ulcers;
* Have taken any prescription drug, over-the-counter drug, vitamin product or herbal medicine within 14 days prior to screening;
* Have taken any drug that inhibit gastric acid secretion, such as H2 receptor antagonist famotidine and proton pump inhibitor omeprazole;
* Have participated in any clinical trial or taken any study drug within 3 months before dosing;
* Positive test result of HBV,HIV or syphilis;
* Solid organ transplanters

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-01-21 (Actual)

PRIMARY OUTCOMES:
Adverse Events,laboratory abnormalities and other abnormalities | 8 days
  Number of participants with Adverse Events, laboratory abnormalities and other abnormalities following dose administration of HEC74647
Antiviral Activity | 8 days
  Change from baseline in HCV RNA following dose administration of HEC74647
Sequence changes in the NS5A coding region | 8 days
  Sequence changes in the NS5A coding region of HCV following multiple dose administration of HEC74647 and for up to 8 days thereafter
Cmax | 8 days
  Maximum observed plasma concentration of HEC74647
Tmax | 8 days
  Time of the maximum observed plasma concentration
AUC | 8 days
  Area under the plasma concentration-time curve (AUC)
t1/2 | 8 days
  Terminal elimination half-life

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Doctor, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- The First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No